CLINICAL TRIAL: NCT04767087
Title: Honey and Nigella Sativa in the Prophylaxis of COVID-19: A Randomized Controlled Trial
Brief Title: Honey and Nigella Sativa in COVID-19 Prophylaxis
Acronym: HNS-COVID-PK
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Registrar Cardiology, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SZMC/IRB/Internal/273/2021
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: Honey; Nigella sativa; Prophylaxis; COVID-19; Prophetic Medicine
MeSH Terms: conditions — COVID-19 | interventions — Honey; Nigella sativa oil

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Honey and Nigella sativa Arm (Active Comparator): 0.5 g/kg/day honey 40 mg/Kg/day Nigella sativa seeds
  Interventions: Drug: Honey; Drug: Nigella sativa seed
- Placebo Arm (Placebo Comparator): empty capsule with sugar water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Honey — 0.5 gm/Kg/day honey
  Arms: Honey and Nigella sativa Arm
Drug: Nigella sativa seed — 40 mg/Kg/day
  Arms: Honey and Nigella sativa Arm
Other: Placebo — empty capsule with sugar water
  Arms: Placebo Arm

SUMMARY:
Honey and Nigella sativa has established antiviral, antibacterial, anti-inflammatory, and immunomodulatory roles. So it is planned to test for its prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals Post-exposure COVID-19

Exclusion Criteria:

* Multi-organ failure active COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection rate | 14 days
  RT-PCR SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Sohaib Ashraf, MBBS, Study Director — Massachusetts General Hospital; Muhammad Ashraf, PhD, Study Chair — University of Veterinary and Animal Sciences; Ahmad Imran, MBBS, Principal Investigator — Shaikh Zayed Post-Graduate Medical Institute; Moneeb Ashraf, MBBS, Principal Investigator — King Edward Medical University
Locations (1):
- Shaikh Zayed Post-Graduate Medical Institute, Lahore, MA, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ashraf S, Ashraf S, Akmal R, Ashraf M, Kalsoom L, Maqsood A, Imran MA, Farooq I, Ashraf S, Siddiqui UN, Ghufran M, Akram MK, Majeed N, Rafique S, Habib Z, Shahab MS, Akmal A, Shaukat Z, Abdin ZU, Khaqan A, Arshad S, Rehman Virk MA, Gul M, Awais AB, Hassan M, Khalid N, Iqbal QUA, Ahmad T, Akram M, Muhammad A, Khalil M, Aslam A, Umer M, Sherazi SSH, Safdar Z, Ahmad S, Bilal M, Zahid MN, Koshak AE, Hilal A, Malik AA, Iqbal U, Baig AA, Alahmadi YM, Humayun A, Malik A, Ahmad A, Ashraf M, Saboor QA, Izhar M; DOCTORS LOUNGE consortium. Prophylactic potential of honey and Nigella sativa L. against hospital and community-based SARS-CoV-2 spread: a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Sep 15;22(1):618. doi: 10.1186/s13063-021-05510-3. PMID 34526081